CLINICAL TRIAL: NCT03190668
Title: Skeletal Muscle and Adipose Tissue Concentrations of Cefazolin Comparing Two Different Dosing Regimens During Pediatric Posterior Spinal Fusion Surgery
Brief Title: Skeletal Muscle and Adipose Tissue Study
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: University of Florida (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: IRB201701129 -A; OCR18899 (Other: University of Florida)
Record Dates: First submitted 2017-06-15; First posted 2017-06-19 (Actual); Results first posted 2023-07-11 (Actual); Last update posted 2023-07-11 (Actual); Status verified 2023-06

CONDITIONS: Idiopathic Scoliosis
Keywords: tissue microdialysis; spinal fusion; surgical site infection
MeSH Terms: conditions — Surgical Wound Infection

STUDY DESIGN:
Intervention Model Description: Simple randomization will be used with each patient has probability 0.5 to be assigned in Group I or Group II. Computer program will generate a uniform random variable between 0 to 1, with subject assigned to Group I if the value is less than 0.5 and assigned to Group II if the value is greater than 0.5.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (2):
- First Regimen Group (Active Comparator): The first regimen will consist of a bolus dose of Cefazolin 30mg/kg up to a maximum of 2000mg IV administered prior to surgical incision. The same pre-operative dose of Cefazolin will be repeated every 3 hours until the completion of surgery. Two will paraspinal muscle microdialysis catheters and two subcutaneous microdialysis catheters will be inserted.
  Interventions: Drug: Bolus dose of Cefazolin; Device: Paraspinal muscle microdialysis catheters; Device: Subcutaneous microdialysis catheters
- Second Regimen Group (Active Comparator): The second regimen will consist of an initial bolus dose of 30 mg/kg up to maximum of 2000 mg. Following the initial bolus dose a continuous Cefazolin drip will start until the end of surgery. Cefazolin drip dose will be 10 mg/(kg*h) up to maximum of 667 mg/h.Two microdialysis catheters will be inserted into a paraspinal muscle and two microdialysis catheters will be inserted subcutaneously.
  Interventions: Drug: Continuous Cefazolin drip; Device: Paraspinal muscle microdialysis catheters; Device: Subcutaneous microdialysis catheters

INTERVENTIONS:
Drug: Bolus dose of Cefazolin — Mode of Cefazolin administration will be a intermittent bolus
  Other Names: Standard mode of prophylactic cefazolin administration
  Arms: First Regimen Group
Drug: Continuous Cefazolin drip — Mode of Cefazolin administration will be a continuous drip
  Other Names: Continuous infusion of prophylactic cefazolin
  Arms: Second Regimen Group
Device: Paraspinal muscle microdialysis catheters — Two dialysis probes will be inserted into a paraspinal muscle
  Other Names: Paraspinal muscle dialysate sample
Device: Subcutaneous microdialysis catheters — Two dialysis probes will be inserted into a paraspinal subcutaneous region
  Other Names: Subcutaneous dialysate sample

SUMMARY:
The purpose of this research study is to compare the current standard of care for prophylactic Cefazolin administered every 3 hours intravenously with continuous infusion of Cefazolin during pediatric spinal surgery.

DETAILED DESCRIPTION:
Determine the skeletal muscle and adipose tissue disposition of prophylactic Cefazolin using microdialysis sampling in a cohort of patients diagnosed with idiopathic scoliosis undergoing posterior spinal fusion (PSF) for administration of Cefazolin by either continuous infusion or intermittent bolus.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of idiopathic scoliosis
* Planned posterior spinal fusion surgery (PSFS)
* Age: 12-20 years old
* American Society of Anesthesiology status I or II undergoing posterior spinal fusion for at least 6 levels
* No known allergy to cefazolin

Exclusion Criteria:

* Known allergy to cefazolin
* Anatomical or other abnormalities that precluded insertion of a microdialysis catheter into the selected paraspinal muscle
* Known renal or hepatic insufficiency or failure

Ages: 12 Years to 20 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 12 (Actual)
Dates: Start 2018-05-29 (Actual); Primary Completion 2022-06-23 (Actual); Study Completion 2022-06-23 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Christoph Seubert, MD, Principal Investigator — University of Florida
Locations (1):
- University of Florida, Gainesville, Florida, United States

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | First Regimen Group | Second Regimen Group
Started | 6 | 6
Completed | 6 | 6
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Population: One subject was withdrawn from each group and not included in the analysis due to insufficient data.
Groups:
- Total: Total of all reporting groups
Arm/Group | First Regimen Group | Second Regimen Group | Total
Number analyzed (Participants) | 6 | 6 | 12
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 6 | 6 | 12
  Between 18 and 65 years | 0 | 0 | 0
  >=65 years | 0 | 0 | 0
Age, Continuous [Mean (Full Range); unit: years] | 15.2 [13 to 17] | 12.8 [12 to 15] | 14 [12 to 17]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 3 | 0 | 3
  Male | 3 | 6 | 9
Race and Ethnicity Not Collected [Count of Participants; unit: Participants] — Population: Race and Ethnicity were not collected from any participant.
Region of Enrollment [Number; unit: participants]
  United States | 6 | 6 | 12

OUTCOME MEASURES:

1. Primary Outcome: Unbound Cefazolin Concentration in Skeletal Muscle
Description: First regimen and second regimen difference between unbound Cefazolin concentrations in the interstitial fluid of skeletal muscle
Time Frame: Changes from baseline (pre-op) up to end of surgical procedure
Measure: Median (75% Confidence Interval); unit: µg/ml/kg
Arm/Group | First Regimen Group | Second Regimen Group
Number analyzed (Participants) | 5 | 5
µg/ml/kg | 3.22 [1.77 to 7.62] | 5.84 [3.01 to 11.35]

2. Primary Outcome: Unbound Cefazolin in Adipose Tissue
Description: First regimen and second regimen difference between unbound Cefazolin concentrations in the interstitial fluid of adipose tissue
Time Frame: Changes from baseline (pre-op) up to end of surgical procedure
Measure: Median (75% Confidence Interval); unit: µg/ml/kg
Arm/Group | First Regimen Group | Second Regimen Group
Number analyzed (Participants) | 5 | 5
µg/ml/kg | 3.21 [2.33 to 8.24] | 6.13 [3.20 to 11.22]

ADVERSE EVENTS:
Time Frame: 1 day
Arm/Group | First Regimen Group | Second Regimen Group
All-Cause Mortality (participants affected / at risk) | 0/6 | 0/6
Serious Adverse Events (participants affected / at risk) | 0/6 | 0/6
Other Adverse Events (participants affected / at risk) | 0/6 | 0/6

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2018-08-27): https://cdn.clinicaltrials.gov/large-docs/68/NCT03190668/Prot_SAP_001.pdf